CLINICAL TRIAL: NCT06658639
Title: Ultrasound Lipolysis Versus Cryolipolysis On Lipid Profile Levels In Centrally Obese Middle Aged Men
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mustafa awad ali awad, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mustafa-004363
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Ultrasound Lipolysis; Cryolipolysis; Lipid Profile; Central Obesity
MeSH Terms: conditions — Obesity, Abdominal | interventions — Caloric Restriction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ultrasound lipolysis group (Experimental): it involves 22 participants and will receive ultrasound lipolysis on abdominal area and low caloric diet treatment. abdominal area was treated for 60-minute session every 2 weeks for 3 months
  Interventions: Device: Ultrasound lipolysis; Other: Low Caloric Diet
- cryolipolysis group (Active Comparator): it involves 22 participants and will receive cryolipolysis on abdominal area and low caloric diet treatment. Each participant underwent a cryolipolysis session on the same abdominal area every 2 weeks for 3 months
  Interventions: Device: Cryolipolysis; Other: Low Caloric Diet
- low caloric diet group (Active Comparator): it involves 22 participants and will receive low caloric diet treatment for 3 months.
  Interventions: Other: Low Caloric Diet

INTERVENTIONS:
Device: Ultrasound lipolysis — Ultrasound lipolysis uses a Luvitra device to emit low-frequency ultrasound pulsed waves. The abdominal area is divided into two sections and the patient is placed in a comfortable supine lying position. The cavitation head is applied slowly to each segment in small circular movements. The treatment lasts 30 minutes on each side, with each session lasting 60 minutes. The same abdominal area is treated every two weeks for three months. The procedure involves cleaning the skin with alcohol cotton.
  Arms: ultrasound lipolysis group
Device: Cryolipolysis — The study utilized Lipocool, a cryolipolysis apparatus from Korea, with a thermoelectric cooling element. Participants were treated with thermal coupling gel on their abdomen, and the tissue was drawn into the applicator with a moderate vacuum. The device was used for 40-50 minutes, with energy extraction controlled by sensors. The system stopped cold exposure and the clinician released the vacuum. Participants underwent cryolipolysis sessions every 2 weeks for 3 months.
  Arms: cryolipolysis group
Other: Low Caloric Diet — A low-calorie diet is a structured plan that restricts daily caloric intake, often used for weight loss. It involves consuming 1,200 to 1,500 calories daily, creating a calorie deficit. However, it requires discipline and safety. The diet is low in fat (20-25%), high in complex carbohydrates (60%), and sufficient in protein (25-50%).

SUMMARY:
The study compares the effects of ultrasound lipolysis and cryo lipolysis on cholesterol, triglyceride, high density lipoprotein, low density lipoprotein, body mass index, skin thickness, waist circumference, and waist hip ratio in centrally obese middle aged men. It also investigates the impact of ultrasound lipolysis on skin thickness, waist circumference, and waist hip ratio.

DETAILED DESCRIPTION:
Obesity has become a key risk factor for the development of cardiovascular diseases and dyslipidemia. Overweight and abdominal obesity has increased in men more than in women.

For young individuals, intra-abdominal fat is the important component of the body fat for six of the eight metabolic risk factors. Intra-abdominal fat might contribute to that most patients with acute myocardial infarction at a young age are men.

Abdominal lipolysis by ultra sonic is a safe and efficacious method and can effectively decrease waist circumference, waist hip ratio and blood cholesterol.

Adding cryolipolysis to a low-calorie diet is protocol from other methods to improve the body profile, in form of body mass index, waist-to-hip ratio, as well subcutaneous fat tissues thickness, but also leads to improvement in lipid profile and liver enzymes

ELIGIBILITY:
Inclusion Criteria:

1. Obese men with middle age range will be 40-60 years.
2. Obese men with central obesity.
3. Body mass index (BMI) greater than 30 Kg \m2.
4. Waist circumference will be >94 cm.
5. Waist to hip ratio more than 0.9

Exclusion Criteria:

1. Chronic respiratory disorders and cardiovascular problems.
2. Diabetic patients.
3. Presence of skin diseases in abdominal regions that prevent the use of ultra sound or cryolipolysis therapy.
4. Men with kidney or liver diseases.
5. Tumor diseases
6. Lesions of higher center leading to obesity.
7. History of active or chronic infectious, autoimmune disease.
8. History of abdominal surgeries.

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 1. Obese men with middle age range will be 40-60 years.
  2. Obese men with central obesity.
  3. Body mass index (BMI) greater than 30 Kg \m2
Enrollment: 66 (Estimated)
Dates: Start 2024-11-05 (Estimated); Primary Completion 2025-03-05 (Estimated); Study Completion 2025-04-05 (Estimated)

PRIMARY OUTCOMES:
assessment of change of lipid profile | at baseline and after 3 months
  A low-calorie diet is a structured plan that restricts daily caloric intake, often used for weight loss. It involves consuming 1,200 to 1,500 calories daily, creating a calorie deficit. However, it requires discipline and safety. The diet is low in fat (20-25%), high in complex carbohydrates (60%), and sufficient in protein (25-50%).

SECONDARY OUTCOMES:
assessment of BMI using Body weight and height scale | at baseline and after 3 months
  For measuring weight in kg and height in cm to calculate the body mass index (BMI) by dividing weight in kg on Height in meter square
assessment of change of skin fold thickness using skin caliper | at baseline and after 3 months
  A caliper is used to measure suprailiac skinfold thickness where subcutaneous fat is pulled away from the muscle with the caliper tongs situated at their ends. For men, the direction of fold pulling was vertical and is taken 2 cm to the side of the umbilicus.
assessment of change of Waist Circumference using tape measurement | at baseline and after 3 months
  A tape, resistant to stretching will be used to measure the waist circumference at the midpoint in line between the lower border of the last felt rib and the iliac crest's highest point. All patients will standing in a comfortable position, with both feet in close proximity, both arms beside the body
assessment of change of Waist Hip Ratio | at baseline and after 3 months
  Using a non-stretchable tape, the hips is measured at the widest part of the hip bones, and the waist is measured at the midpoint in line between the lower border of the last felt rib and the iliac crest's highest point then the WHR will calculated by dividing the waist measurement by the hip measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- out-patient clinic, faculty of physical therapy, Cairo university, Giza, Egypt